CLINICAL TRIAL: NCT05384379
Title: Clinical Study to Evaluate the Efficacy and Safety od BZ371B in Patients With Acute Respiratory Distress System (ARDS) in Mechanical Ventilation, Due to Respiratory Infections
Brief Title: Efficacy and Safety Evaluation of BZ371B in ARDS Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Suboptimal enrollment
Sponsor: Biozeus Biopharmaceutical S.A. (Industry)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZ371CLI301
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: ARDS; ARDS, Human; Pulmonary Disease
Keywords: ARDS; Acute respiratory distress syndrome; Intubation; intubated; critical care; Nitric Oxide; NO; NOS; Nitric Oxide Synthase; BZ371B
MeSH Terms: conditions — Respiratory Distress Syndrome; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated Group (Experimental): Intubated patients treated with inhaled BZ371B will receive a dose of 12 mg of BZ371B divided in two different nebulizations per day, for three cosnecutive days
  Interventions: Drug: Inhaled BZ371B

INTERVENTIONS:
Drug: Inhaled BZ371B — Intubated patients suffering from ARDS will receive BZ371B in a dose of 12 mg. This will be divided into 2 nebulizations, each with 10 ml. The first nebulization is at a dose of 3 mg and the second at a dose of 9 mg.

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and efficacy of BZ371B in intubated patients with severe Acute Respiratory Distress Syndrome.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a severe medical condition that is triggered by an alveolar capillary membrane damage resulted from several causes. Among these causes, respiratory viral infections such as SARS-CoV-2 can be responsible for the development of the disease. ARDS presents a high mortality rate, which may range from 33-52%. The main difficulty for the treatment of this disease is dealing with hypoxia.

Nitric Oxide inhalation therapy has proven to increase oxygenation and Ventilation/Perfusion by it's vasodilation property. However, there are several limitations for it's use, such as the need of a specialized equipment, systemic side effects, etc. The use of others vasodilation medications are not indicated due to their systemic systemic exposure and non-selective vasodilation.

BZ371B is a small peptide that acts as a NO synthase (NOS) enhancer, inducing local NO production, and is capable to present local vasodilation effect increasing blood flow regulation, by a new and innovative mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Men or Women
* In Mechanical Ventilation
* Diagnosed with Acute Respiratory Dystress Syndrome characterized by: acute beginning (less than one week from the beggining of the disease); bilateral opacity in the Torax X-Ray (not explained by stroke, atelectasis or nodules); respiratory failure not derived from cardiac failure and water overload.
* P/F lower or equal to 150 mmHg with FiO2 higher or equal to 70% and PEEP higher or or equal to 88 mmHg
* ALready executed first pronation, followed by supine position. One hour after returning from supine position.

Exclusion Criteria:

* Presence of pulmonary thromboembolism
* Presence of secondary bacterial pneumonia
* Severe Asthma
* Pregnant or lactanting women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
P/F ratio | 4 days
  PaO2 divided by FiO2 measurement
Shunt ratio | 4 days
  Shunt ratio measurement
Ventilation-Perfusion (V/Q) ratio | 4 days
  V/Q measurement
Systemic blood pressure (SBP) | 4 days
  SBP measurement
Cardiac Function | 4 days
  Heart Rate (HR) and Ejection Fraction measurement
Adverse Effect | 4 days
  Adverse effect evaluation of compound use and application

SECONDARY OUTCOMES:
Pulmonary arterial pressure (PAP) | 4 days
  PAP measurement
Pulmonary vascular resistence | 4 days
  Pulmonary vascular resistance measurement

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP Amato, Phd, Principal Investigator — Department of Cardio-Pulmonar, Pulmonary Division, Hospital das Clínicas, University of São Paulo
Locations (1):
- InCor USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No